CLINICAL TRIAL: NCT01424124
Title: Randomized, Double-blind, Placebo/Active-controlled, Multi-center Clinical Trial to Investigate the Safety/Tolerability and Efficacy of YHD001 Following 8 Weeks Oral Administration of YHD001 in Patients With Partially Controlled Asthma
Brief Title: Safety and Efficacy of YHD001 in Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YHD001-201
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- YHD001 dose level 1 (Experimental)
  Interventions: Drug: YHD001 dose level 1
- YHD001 dose level 2 (Experimental)
  Interventions: Drug: YHD001 dose level 2
- Singulair (Active Comparator)
  Interventions: Drug: Singulair
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YHD001 dose level 1 — Tablet, three times daily / 8 weeks
  Arms: YHD001 dose level 1
Drug: YHD001 dose level 2 — Tablet, three times daily / 8 weeks
  Arms: YHD001 dose level 2
Drug: Singulair — Tablet, one times daily / 8 weeks
  Arms: Singulair
Drug: Placebo — Tablet, one times daily / 7 days
  Arms: Placebo

SUMMARY:
The main objective is to evaluate the safety/tolerability and efficacy of YHD001 compared to singulair or placebo in patients (n=96) with partially controlled asthma.

The study will conduct with 4 comparative groups orally treated with YHD001 dose level 1(t.i.d.), YHD001 dose level 2(t.i.d.), singulair 10mg(q.d.) or Placebo for 8 weeks.

DETAILED DESCRIPTION:
Singulair: Montelukast sodium (leukotriene modulator)

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent
* Acceptable medical history, physical exam,laboratory tests and EKG, during screening
* Nonsmoking (for longer than 1 year) patients with asthma
* Reversible airways obstruction (an increase in FEV1 absolute value of 12% or greater) 20 to 30 minutes after inhalation of b-agonist
* FEV1 between 50% and 85% of the predicted value (withholding short-acting, inhaled b2-adrenergic agonist for 6 hours)

Exclusion Criteria:

* History of any clinically significant disease
* History of drug/chemical/alcohol abuse
* Active upper respiratory tract infection within 3 weeks, emergency room treatment for asthma within 1 month, or hospitalization for asthma within 3 months of the prestudy visit

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline of FEV1 at week 4 | Baseline, week 4
  FEV1: Forced Expiratory Volume In One Second

SECONDARY OUTCOMES:
Change from baseline of FEV1 at week 8 | Baseline, week 8
Change from baseline of PEFR at week 8 | Baseline, week 8
  PEFR: Peak Expiratory Flow Rate
Change from baseline of ACT Score at week 8 | Baseline, week 8
  ACT: Asthma control test
Change from baseline of using rescue medication(b-Agonist) at week 8 | Baseline, week 8
safety assessment | week 9
  Comparison of the adverse event profiles throughout the course of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea